CLINICAL TRIAL: NCT00055497
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study of the Human Anti-TNF Monoclonal Antibody Adalimumab for the Maintenance of Clinical Remission in Subjects With Crohn's Disease
Brief Title: Remission in Subjects With Crohn's Disease, 1 Year Phase
Acronym: CLASSICII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Anne Camez, Medical Director, Abbott
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M02-433
Record Dates: First submitted 2003-03-03; First posted 2003-03-05 (Estimated); Results first posted 2010-05-18 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Double-Blind Method; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Double-blind (DB) adalimumab placebo (Placebo Comparator): Double-blind nonactive matching subcutaneous injection
  Interventions: Biological: Double-blind (DB) adalimumab placebo
- Double-blind adalimumab 40 mg every other week (eow) (Experimental): Double-blind adalimumab 40 mg eow by subcutaneous injection
  Interventions: Biological: DB adalimumab 40 mg eow
- Double-blind adalimumab 40 mg every week (ew) (Experimental): Double-blind adalimumab 40 mg every week by subcutaneous injection
  Interventions: Biological: DB adalimumab 40 mg ew
- Open-label adalimumab 40 mg (Experimental): Open-label adalimumab 40 mg eow or ew by subcutaneous injection
  Interventions: Biological: OL adalimumab 40 mg

INTERVENTIONS:
Biological: Double-blind (DB) adalimumab placebo — Double-blind nonactive matching subcutaneous injection
  Other Names: Humira®
  Arms: Double-blind (DB) adalimumab placebo
Biological: DB adalimumab 40 mg eow — Double-blind adalimumab 40 mg every other week by subcutaneous injection
  Other Names: Humira®
  Arms: Double-blind adalimumab 40 mg every other week (eow)
Biological: DB adalimumab 40 mg ew — Double-blind adalimumab 40 mg every week by subcutaneous injection
  Other Names: Humira®
  Arms: Double-blind adalimumab 40 mg every week (ew)
Biological: OL adalimumab 40 mg — Open-label adalimumab every other week or every week by subcutaneous injection
  Other Names: Humira®
  Arms: Open-label adalimumab 40 mg

SUMMARY:
The objectives were: (1) To demonstrate the efficacy of adalimumab in the maintenance of clinical remission up to 56 weeks in participants with Crohn's disease who participated in NCT00055523; (2) To delineate the safety of adalimumab when administered to participants with Crohn's disease up to 56 weeks.

DETAILED DESCRIPTION:
Study NCT00055497 was designed to evaluate the efficacy and safety of adalimumab in the maintenance of clinical remission in patients with Crohn's disease (CD). The study consisted of 2 phases: 1. the first year phase lasting until Week 56 and consisting of a randomized, double-blind (DB), placebo-controlled portion (NCT00055497) and of a concomitant open label (OL) portion, and 2. a long-term extension phase (NCT01070303) that lasted 264 additional weeks (Week 56 to Week 320).

Potential participants were screened at the time of enrollment in the lead-in, induction therapy study (NCT00055523). Participants who completed the lead-in study, NCT00055523, were eligible to participate in the rollover study, NCT00055497.

In Study NCT00055497, all participants received 40 mg of adalimumab subcutaneously (SC) at Baseline (Week 0) and Week 2 of Study NCT00055497. Baseline of Study NCT00055497 is synonymous with NCT00055523 Week 4. At Week 4 of Study NCT00055497, participants were randomized based on their clinical remission status at Baseline and Week 4 of Study NCT00055497. Participants who demonstrated clinical remission (defined as a Crohn's Disease Activity Index [CDAI] score < 150 points) at Baseline of Study NCT00055497 and who remained in clinical remission at Week 4 of Study NCT00055497 (those participants constituted the randomized analysis set) were randomized to receive 1 of 3 blinded treatments: adalimumab 40 mg every other week (eow), adalimumab 40 mg every week (ew), or placebo. Participants who did not demonstrate clinical remission at Baseline of Study NCT00055497, or who were no longer in clinical remission at Week 4 of Study NCT00055497 were assigned to receive OL adalimumab 40 mg eow; those participants constituted the OL analysis set. At any time during Study NCT00055497, participants receiving OL adalimumab 40 mg SC eow who developed a flare or were non-responders during OL treatment could have had his/her dose increased to 40 mg SC weekly. Participants who were documented as having completed Week 56 are counted in the study completion total.

After 1 year (Week 56), participants who met eligibility criteria for the long-term extension phase (NCT01070303) were switched to OL adalimumab 40 mg subcutaneous (SC) eow, and participants previously in the OL treatment group of Study NCT00055497 continued on their previous OL adalimumab dose (adalimumab 40 mg SC eow or every week).

ELIGIBILITY:
Inclusion:

* Patient must have successfully completed the induction study NCT00055523
* Diagnosis of Crohn's disease
* Willing and able to give informed consent

Exclusion:

* Diagnosis of ulcerative colitis
* Pregnancy or breastfeeding
* Previous use of infliximab or other anti-TNF antagonists
* Previous history of active tuberculosis or listeria infection
* Previous history of cancer other than successfully treated skin cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2002-08; Primary Completion 2005-01 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Camez, MD, Study Director — Abbott
Locations (43):
- United States (43):
  - Gastroenterology Associates of the East Bay, Berkeley, California
  - Long Beach Gastroenterology Assoc., Long Beach, California
  - Sharp Rees-Stealy Medical Group, San Diego, California
  - Gastroenterology Assoc. of Fairfield Co., Bridgeport, Connecticut
  - Cleveland Clinic Florida, Weston, Florida
  - Wake Research Associates, Weston, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Atlanta Gastroenterology Assoc., Atlanta, Georgia
  - Southeastern Digestive & Liver Disease, Savannah, Georgia
  - Northwest Gastroenterologists, S.C., Arlington Heights, Illinois
  - University of Chicago, Chicago, Illinois
  - Drug Research Services, Inc., Metairie, Louisiana
  - LSU School of Medicine, New Orleans, Louisiana
  - Digestive Disorders Associates, Annapolis, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Clinical Pharmacology Study Group, Worchester, Massachusetts
  - Mayo Clinic and Mayo Foundation, Rochester, Minnesota
  - Gastroenterology and Hepatology, Kansas City, Missouri
  - Glenn Gordon, MD, Mexico, Missouri
  - Deaconess Billings Clinic Research Division, Billings, Montana
  - Gastroenterology Specialties, P.C., Lincoln, Nebraska
  - Long Island Clinical Research Associates, Great Neck, New York
  - NY Center for Clinical Research, Lake Success, New York
  - New York Presbyterian Hospital, New York, New York
  - Daniel Present, New York, New York
  - Rochester Institute for Digestive Diseases, Rochester, New York
  - UNC School of Medicine, Chapel Hill, North Carolina
  - Charlotte Gastroenterology and Hepatology, Charlotte, North Carolina
  - Carolina Research Associates, Charlotte, North Carolina
  - Digestive Health Specialists, Winston-Salem, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Oklahoma Foundation for Digestive Disease, Oklahoma City, Oklahoma
  - Research Solutions, Tulsa, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Peter Molloy, MD, Pittsburgh, Pennsylvania
  - Diseases of the Digestive System, Chattanooga, Tennessee
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Northwest Gastroenterology, Bellevue, Washington
  - Inland Empire Gastroenterology, Spokane, Washington
  - Tacoma Digestive Disease Center, Tacoma, Washington
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Ryan C, Sobell JM, Leonardi CL, Lynde CW, Karunaratne M, Valdecantos WC, Hendrickson BA. Safety of Adalimumab Dosed Every Week and Every Other Week: Focus on Patients with Hidradenitis Suppurativa or Psoriasis. Am J Clin Dermatol. 2018 Jun;19(3):437-447. doi: 10.1007/s40257-017-0341-6. PMID 29380251
- [Derived] Steenholdt C, Al-khalaf M, Brynskov J, Bendtzen K, Thomsen OO, Ainsworth MA. Clinical implications of variations in anti-infliximab antibody levels in patients with inflammatory bowel disease. Inflamm Bowel Dis. 2012 Dec;18(12):2209-17. doi: 10.1002/ibd.22910. Epub 2012 Feb 16. PMID 22344964

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 276 participants were enrolled in the present study from 53 sites in the United States (US), Canada, Poland, Belgium, the Netherlands, and Czech Republic. The first visit in the present study for the first participant was 28 August 2002 and the final visit for the last participant occurred on 12 January 2005.
Pre-assignment Details: Study was rollover of NCT00055523; screening done in NCT00055523. At Week 4 of NCT00055497, 55 remitters at Week 0 and Week 4 of Study NCT00055497 were randomized to DB therapy; 204 non-remitters were assigned to OL adalimumab. 17 discontinued before/at Week 4, included in OL group for Participant Flow and AEs because they were not randomized.
Groups:
- DB Placebo: Double-blind adalimumab placebo every week.
- DB Adalimumab 40 mg Every Other Week (Eow): Double-blind adalimumab 40 mg every other week (injection received every week; placebo received when active drug not received)
- DB Adalimumab 40 mg Every Week (ew): Double-blind adalimumab 40 mg every week.
- OL Adalimumab 40 mg: Open-label adalimumab 40 mg every other week or every week.
Period: Overall Study
Arm/Group | DB Placebo | DB Adalimumab 40 mg Every Other Week (Eow) | DB Adalimumab 40 mg Every Week (ew) | OL Adalimumab 40 mg
Started | 18 | 19 | 18 | 221 (17 participants who discontinued at/before Week 4 are counted here because they were not randomized.)
Completed | 13 (Participants may have continued to the open-label extension study. See NCT01070303.) | 16 (Participants may have continued to the open-label extension study. See NCT01070303.) | 16 (Participants may have continued to the open-label extension study. See NCT01070303.) | 131 (Participants may have continued to the open-label extension study. See NCT01070303.)
Not Completed | 5 | 3 | 2 | 90
Not completed — Adverse Event | 1 | 1 | 1 | 28
Not completed — Withdrawal by Subject | 3 | 1 | 1 | 15
Not completed — Lost to Follow-up | 0 | 1 | 0 | 5
Not completed — Protocol Violation | 0 | 0 | 0 | 3
Not completed — Lack of Efficacy | 1 | 0 | 0 | 27
Not completed — Administrative Reasons | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 11

BASELINE CHARACTERISTICS:
Groups:
- OL Adalimumab 40 mg Eow: Participants who did not continue at Week 4 are not included in Baseline summary.
- Total: Total of all reporting groups
Arm/Group | DB Placebo | DB Adalimumab 40 mg Every Other Week (Eow) | DB Adalimumab 40 mg Every Week | OL Adalimumab 40 mg Eow | Total
Number analyzed (Participants) | 18 | 19 | 18 | 204 | 259
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 1 | 1
  Between 18 and 65 years | 17 | 19 | 18 | 195 | 249
  >=65 years | 1 | 0 | 0 | 8 | 9
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline data were collected in the lead-in study (NCT00055523) and are reported by treatment group determined at Week 4 of NCT00055497.
  Participants
    Female | 12 | 12 | 9 | 104 | 137
    Male | 6 | 7 | 9 | 100 | 122

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants Achieving Clinical Remission at Week 24 - NRI
Description: Clinical remission is defined as CDAI score <150. CDAI evaluates 8 Crohn's-related variables during a 1-week assessment period, yielding a composite score >/= 0 and without upper limit. The range of scores during Study NCT00055497 and the lead-in study (NCT00055523) was 0 to 633. A lower score indicates less severe Crohn's disease activity.
Time Frame: Week 24
Population: Participants randomized to DB treatment who received at least one injection of blinded study drug were included in assigned treatment group. Participants in the OL adalimumab group were all participants who were assigned to the OL treatment and continued past Week 4. Nonresponder imputation (NRI) (CR-100 not achieved) was used for missing data.
Measure: Number; unit: Participants
Arm/Group | DB Placebo | DB Adalimumab 40 mg Every Other Week (Eow) | DB Adalimumab 40 mg Every Week (ew) | OL Adalimumab 40 mg Eow
Number analyzed (Participants) | 18 | 19 | 18 | 204
Participants | 7 | 11 | 17 | 74

2. Secondary Outcome: Number of OL Participants Achieving Clinical Remission at Week 56 - NRI
Description: as for outcome 1
Time Frame: Week 56
Population: Participants in the OL adalimumab group were all participants who were assigned to the OL treatment and continued past Week 4. Nonresponder imputation (NRI) (CR-100 not achieved) was used for missing data.
Measure: Number; unit: Participants
Arm/Group | OL Adalimumab 40 mg
Number analyzed (Participants) | 204
Participants | 74

3. Primary Outcome: Number of Randomized Participants Achieving Clinical Remission at Week 56 - Non-Responder Imputation (NRI)
Description: as for outcome 1
Time Frame: Week 56
Population: Participants randomized to DB treatment who received at least one injection of blinded study drug were included in assigned treatment group. Nonresponder imputation (NRI) (clinical remission not achieved) was used for missing data.
Measure: Number; unit: Participants
Arm/Group | Placebo | DB Adalimumab 40 mg Every Other Week (Eow) | DB Adalimumab 40 mg Every Week (ew)
Number analyzed (Participants) | 18 | 19 | 18
Participants | 6 | 9 | 12
Statistical Analysis 1: Comparison: Placebo vs DB Adalimumab 40 mg Every Other Week (Eow) vs DB Adalimumab 40 mg Every Week (ew); Test type: Superiority or Other; p = 0.142, Log Rank

4. Primary Outcome: Number of Randomized Participants Achieving Clinical Remission at Week 56 - Last Observation Carried Forward (LOCF)
Description: as for outcome 1
Time Frame: Week 56
Population: Participants randomized to DB treatment who received at least one injection of blinded study drug were included in assigned treatment group. Last observation carried forward was used for missing data.
Measure: Number; unit: Participants
Arm/Group | DB Placebo | DB Adalimumab 40 mg Every Other Week (Eow) | DB Adalimumab 40 mg Every Week (ew)
Number analyzed (Participants) | 18 | 19 | 18
Participants
  Week 56 | 8 | 15 | 15
Statistical Analysis 1: Comparison: DB Placebo vs DB Adalimumab 40 mg Every Other Week (Eow) vs DB Adalimumab 40 mg Every Week (ew); Test type: Superiority or Other; p = 0.029, Fisher Exact

5. Secondary Outcome: Number of Participants Achieving Clinical Response 100 (CR-100) - NRI
Description: A CR-100 is a decrease from Baseline of lead-in study (NCT00055523) in CDAI score of 100 or more points, indicating significant improvement in disease severity. CDAI evaluates 8 Crohn's-related variables during a 1-week assessment period, yielding a composite score >/= 0 and without upper limit. The range of scores during Study NCT00055497 and the lead-in study (NCT00055523) was 0 to 633. A lower score indicates less severe Crohn's disease activity.
Time Frame: From Baseline of lead-in study to Week 24 and Week 56
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | DB Placebo | DB Adalimumab 40 mg Eow | DB Adalimumab 40 mg ew | OL Adalimumab 40 mg Eow
Number analyzed (Participants) | 18 | 19 | 18 | 204
Participants
  Week 24 | 7 | 11 | 17 | 110
  Week 56 | 6 | 9 | 13 | 101
Statistical Analysis 1: Comparison: DB Placebo vs DB Adalimumab 40 mg Eow; Week 24; Test type: Superiority or Other; p = 0.330, Fisher Exact
Statistical Analysis 2: Comparison: DB Placebo vs DB Adalimumab 40 mg ew; Week 24; Test type: Superiority or Other; p = 0.001, Fisher Exact
Statistical Analysis 3: Comparison: DB Placebo vs DB Adalimumab 40 mg Eow; Week 56; Test type: Superiority or Other; p = 0.508, Fisher Exact
Statistical Analysis 4: Comparison: DB Placebo vs DB Adalimumab 40 mg ew; Week 56; Test type: Superiority or Other; p = 0.044, Fisher Exact

6. Secondary Outcome: Number of Participants Achieving Clinical Response 70 (CR-70)- NRI
Description: A CR-70 is a decrease from Baseline of lead-in study (NCT00055523) in CDAI score of 70 or more points, indicating a significant improvement in disease severity. CDAI evaluates 8 Crohn's-related variables during a 1-week assessment period, yielding a composite score >/= 0 and without upper limit. The range of scores during Study NCT00055497 and the lead-in study (NCT00055523) was 0 to 633. A lower score indicates less severe Crohn's disease activity.
Time Frame: From Baseline of lead-in study to Week 24 and to Week 56
Population: Participants randomized to DB treatment who received at least one injection of blinded study drug were included in assigned treatment group. Participants in the OL adalimumab group were all participants who were assigned to the OL treatment and continued past Week 4. Nonresponder imputation (NRI) (CR-70 not achieved) was used for missing data.
Measure: Number; unit: Participants
Arm/Group | DB Placebo | DB Adalimumab 40 mg Eow | DB Adalimumab 40 mg ew | OL Adalimumab 40 mg Eow
Number analyzed (Participants) | 18 | 19 | 18 | 204
Participants
  Week 24 | 8 | 13 | 17 | 123
  Week 56 | 6 | 9 | 13 | 110
Statistical Analysis 1: Comparison: DB Placebo vs DB Adalimumab 40 mg Eow; Week 24; Test type: Superiority or Other; p = 0.191, Fisher Exact
Statistical Analysis 2: Comparison: DB Placebo vs DB Adalimumab 40 mg ew; Week 24; Test type: Superiority or Other; p = 0.003, Fisher Exact
Statistical Analysis 3: Comparison: DB Placebo vs DB Adalimumab 40 mg Eow; Week 56; Test type: Superiority or Other; p = 0.508, Fisher Exact
Statistical Analysis 4: Comparison: DB Placebo vs DB Adalimumab 40 mg ew; Week 56; Test type: Superiority or Other; p = 0.004, Fisher Exact

7. Secondary Outcome: Number of Participants Achieving Clinical Remission at Week 24 - LOCF
Description: as for outcome 1
Time Frame: Week 24
Population: Participants randomized to DB treatment who received at least one injection of blinded study drug were included in assigned treatment group. Participants in the OL adalimumab group were all participants who were assigned to the OL treatment and continued past Week 4. Last observation carried forward (LOCF) was used for missing data.
Measure: Number; unit: Participants
Arm/Group | DB Placebo | DB Adalimumab 40 mg Every Other Week (Eow) | DB Adalimumab 40 mg Every Week (ew) | OL Adalimumab 40 mg Eow
Number analyzed (Participants) | 18 | 19 | 18 | 204
Participants
  Week 24 | 7 | 11 | 17 | 82
Statistical Analysis 1: Comparison: DB Placebo vs DB Adalimumab 40 mg Every Other Week (Eow) vs DB Adalimumab 40 mg Every Week (ew); Test type: Superiority or Other; p = 0.001, Fisher Exact

8. Secondary Outcome: Number of OL Participants Achieving Clinical Remission at Week 56 - LOCF
Description: as for outcome 1
Time Frame: Week 56
Measure: Number; unit: Participants
Arm/Group | OL Adalimumab 40 mg
Number analyzed (Participants) | 204
Participants | 93

9. Secondary Outcome: Number of Participants Achieving CR-100 - LOCF
Description: as for outcome 5
Time Frame: From Baseline of lead-in study to Week 24 and Week 56
Population: Subjects randomized to DB treatment who received at least one injection of blinded study drug were included in assigned treatment group. Subjects in the OL adalimumab group were all subjects who were assigned to the OL treatment and continued past Week 4. LOCF was used for missing data.
Measure: Number; unit: Participants
Arm/Group | DB Placebo | DB Adalimumab 40 mg Every Other Week (Eow) | DB Adalimumab 40 mg Every Week (ew) | OL Adalimumab 40 mg Eow
Number analyzed (Participants) | 18 | 19 | 18 | 204
Participants
  Week 24 | 7 | 11 | 17 | 110
  Week 56 | 6 | 9 | 13 | 101

10. Secondary Outcome: Number of Participants Achieving CR-70 - LOCF
Description: as for outcome 6
Time Frame: From Baseline of lead-in study to Week 24 and Week 56
Population: Subjects randomized to DB treatment who received at least one injection of blinded study drug were included in assigned treatment group. Subjects in the OL adalimumab group were all subjects who were assigned to the OL treatment and continued past Week 4. LOCF imputation was used for missing data.
Measure: Number; unit: Participants
Arm/Group | DB Placebo | DB Adalimumab 40 mg Every Other Week (Eow) | DB Adalimumab 40 mg Every Week (ew) | OL Adalimumab 40 mg Eow
Number analyzed (Participants) | 18 | 19 | 18 | 204
Participants
  Week 24 | 15 | 18 | 17 | 144
  Week 56 | 13 | 15 | 16 | 147

11. Secondary Outcome: Change in Inflammatory Bowel Disease Questionnaire (IBDQ) Scores - LOCF
Description: IBDQ is a validated disease-specific instrument that assesses the impact of IBD on patient quality of life during a 2-week recall period. It has 32 questions about bowel function and related symptoms, and their social and emotional impact. For each question, participants selected 1 of 7 responses, where 1=poor quality of life (e.g., feeling of fatigue "all of the time") and 7=good quality on the item (e.g., feeling of fatigue "none of the time"). IBDQ scores range from 32 to 224. Higher scores indicate better quality of life, and increases in IBDQ indicate improved overall quality of life.
Time Frame: Change from Baseline of lead-in study to Week 24 and Week 56
Population: Participants randomized to DB treatment who received at least one injection of blinded study drug were included in assigned treatment group. OL adalimumab group was all participants assigned to the OL treatment who continued past Week 4. LOCF was used for missing data. 4 participants in OL group did not have IBDQ data at Baseline of lead-in study.
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | DB Placebo | DB Adalimumab 40 mg Every Other Week (Eow) | DB Adalimumab 40 mg Every Week (ew) | OL Adalimumab 40 mg Eow
Number analyzed (Participants) | 18 | 19 | 18 | 200
Scores on a scale
  Week 24 | 29.9 [11.0 to 48.9] | 43.4 [27.7 to 59.2] | 51.9 [30.8 to 73.0] | 33.9 [29.7 to 38.1]
  Week 56 | 24.7 [0.7 to 48.7] | 45.7 [27.1 to 64.4] | 45.2 [23.1 to 67.4] | 36.0 [31.3 to 40.6]

ADVERSE EVENTS:
Time Frame: Safety was measured from the first dose of adalimumab, which could have occurred in the lead-in study, NCT00055523, or in NCT00055497 for participants randomized to placebo in the lead-in study.
Description: Events were summarized from Week 0 of NCT00055523, for participants who entered NCT00055497, to Week 56 of NCT00055497. Treatment-emergent AEs=(1) AEs that began on/after 1st study drug dose in Study NCT00055497 and within 70 days after last dose; or (2) increased severity of ongoing AEs that began on/after 1st study drug dose in Study NCT00055523.
Arm/Group | DB Placebo | DB Adalimumab 40 mg Eow | DB Adalimumab 40 mg ew | OL Adalimumab 40 mg
Serious Adverse Events (participants affected / at risk) | 2/18 | 1/19 | 0/18 | 37/221
Other Adverse Events (participants affected / at risk) | 18/18 | 15/19 | 14/18 | 190/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB Placebo (N=18) | DB Adalimumab 40 mg Eow (N=19) | DB Adalimumab 40 mg ew (N=18) | OL Adalimumab 40 mg (N=221)
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 2
Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Abscess intestinal (Infections and infestations) | 0 | 0 | 0 | 1
Anemia NOS aggravated (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Calculus renal (Renal and urinary disorders) | 0 | 0 | 0 | 1
Cerebrovascular accident (Vascular disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 9
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Diverticulitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dizziness (excl vertigo) (Nervous system disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
Fifth disease (Infections and infestations) | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Ileal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc herniation (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intestinal stenosis NOS (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Meningitis viral (Infections and infestations) | 0 | 0 | 0 | 1
Nocardiosis (Infections and infestations) | 0 | 0 | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 2
Pain (General disorders) | 0 | 0 | 0 | 1
Pyloric stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1
Retroperitoneal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 3
Small intestinal stricture (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Sweating increased (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB Placebo (N=18) | DB Adalimumab 40 mg Eow (N=19) | DB Adalimumab 40 mg ew (N=18) | OL Adalimumab 40 mg (N=221)
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 9
Abdominal pain aggravated (Gastrointestinal disorders) | 1 | 0 | 0 | 7
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 3
Abdominal tenderness (Gastrointestinal disorders) | 2 | 2 | 0 | 15
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 10
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Anxiety aggravated (Psychiatric disorders) | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 27
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 14
Chest tightness aggravated (General disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 1 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 8
Crohn's disease aggravated (Gastrointestinal disorders) | 5 | 4 | 2 | 39
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 10
Dizziness (excl vertigo) (Nervous system disorders) | 1 | 1 | 2 | 7
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 1 | 11
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 7
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 4
Fatigue (General disorders) | 2 | 1 | 1 | 16
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Headache (Nervous system disorders) | 2 | 0 | 0 | 31
Influenza (Infections and infestations) | 1 | 3 | 1 | 14
Injection site oedema (General disorders) | 1 | 0 | 0 | 2
Injection site reaction (General disorders) | 1 | 1 | 0 | 11
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 12
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2 | 0 | 8
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 7
Nasopharyngitis (Infections and infestations) | 7 | 5 | 2 | 37
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 23
Pharyngolaryngeal pain (Gastrointestinal disorders) | 2 | 2 | 0 | 11
Pain in limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 11
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 5
Pyrexia (General disorders) | 1 | 1 | 0 | 21
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 15
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 14
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 5
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2 | 19
Urinary tract infection (Infections and infestations) | 2 | 0 | 1 | 13
Viral infection (Infections and infestations) | 0 | 4 | 0 | 6
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 15
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 5
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 2
Conjunctivitis (Eye disorders) | 2 | 0 | 0 | 9
Episcleritis (Eye disorders) | 1 | 0 | 0 | 0
Iritis (Eye disorders) | 0 | 0 | 1 | 1
Pterygium (Eye disorders) | 0 | 0 | 1 | 0
Vision abnormal (Eye disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 0 | 20
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Anal skin tags (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Faecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 3
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 5
Oesophageal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Tooth impacted (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Adverse drug reaction (General disorders) | 1 | 0 | 0 | 2
Application site pain (General disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0
Axillary mass (General disorders) | 0 | 1 | 0 | 0
Bloody drainage (General disorders) | 1 | 0 | 0 | 0
Fall (General disorders) | 1 | 0 | 0 | 3
Fatigue aggravated (General disorders) | 1 | 1 | 0 | 2
Ill-defined disorder (General disorders) | 1 | 0 | 1 | 0
Influenza like illness (General disorders) | 2 | 0 | 0 | 9
Malaise (General disorders) | 0 | 1 | 0 | 2
Oedema (General disorders) | 0 | 1 | 0 | 5
Pain (General disorders) | 2 | 0 | 0 | 6
Tenderness (General disorders) | 0 | 1 | 0 | 4
Abscess (Infections and infestations) | 0 | 1 | 0 | 3
Arthropod infestation (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis acute (Infections and infestations) | 0 | 1 | 0 | 5
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 1
Dry socket (Infections and infestations) | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 1 | 4
Ear infection (Infections and infestations) | 1 | 1 | 0 | 2
Fungal infection (Infections and infestations) | 1 | 1 | 0 | 6
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 8
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 1
Otitis media (Infections and infestations) | 1 | 0 | 0 | 2
Pathogen resistance (Infections and infestations) | 1 | 0 | 0 | 0
Perineal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 1 | 0 | 2
Sinusitis (Infections and infestations) | 1 | 4 | 1 | 20
Vaginal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Vaginal candidiasis (Infections and infestations) | 1 | 0 | 0 | 2
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Abrasion (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 3
Accident (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2
Muscle strain (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Antinuclear factor positive (Investigations) | 2 | 1 | 0 | 5
Blood creatine phophokinase increased (Investigations) | 0 | 0 | 1 | 4
Double-stranded DNA antibody (Investigations) | 0 | 1 | 0 | 1
Eosinophil count increased (Investigations) | 1 | 0 | 0 | 0
Liver function tests abnormal (Investigations) | 1 | 0 | 0 | 1
Lymphocyte morphology abnormal (Investigations) | 0 | 1 | 0 | 0
Monocyte count increased (Investigations) | 1 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 1 | 0 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0
Arthritis enteropathic (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 4
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Polyarthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Sciatica aggravated (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Temporomandibular joint disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Diabetes mellitus aggravated (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Dystrophic calcification (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Hypercholesterolaemia aggravated (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Headache aggravated (Nervous system disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 4
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 1
Sleep apnoea syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Acute stress disorder (Psychiatric disorders) | 0 | 0 | 1 | 3
Adjustment disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 5
Insomnia exacerbated (Psychiatric disorders) | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 1 | 0
Difficulty in micturition (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 7
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Nipple pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3
Chronic obstructive airways disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal passage irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 4
Acrochordons (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 5
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 3
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Skin desquamation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin nodule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2
Continuous positive airway pressure (Surgical and medical procedures) | 0 | 1 | 0 | 0
Endodontic procedure (Surgical and medical procedures) | 0 | 0 | 1 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0 | 1
Vasectomy (Surgical and medical procedures) | 0 | 0 | 1 | 0
Ecchymosis (Vascular disorders) | 1 | 0 | 0 | 3
Petechiae (Vascular disorders) | 0 | 0 | 1 | 0
Mass (General disorders) | 0 | 1 | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 1 | 0 | 3
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 4
Pharyngitis (Infections and infestations) | 2 | 1 | 0 | 3
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.